CLINICAL TRIAL: NCT06355791
Title: The Stability Study: Open-Label, Multi-Center, Post-Market Study of Functional Motion Outcomes In Subjects Treated With the Spinal Simplicity Minuteman G5 Fusion Plate
Brief Title: Post-Market Clinical Study of Functional Motion Outcomes in Subjects Treated With the Minuteman Device
Acronym: STABILITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Simplicity LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDPROJ-4-TP-001-23
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Degenerative Conditions of the Lumbar Spine; Lumbar Spinal Stenosis; Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surgical Group (Other): patient treated with Minuteman G5 interspinous fusion device 510k cleared for degenerative conditions of the lumbar spine
  Interventions: Device: Minuteman G5 Device

INTERVENTIONS:
Device: Minuteman G5 Device — The Minuteman G5 MIS Fusion Plate consists of spinous process plates and surgical instruments. Implants are made of Titanium alloy

SUMMARY:
This is a prospective, multi-center open-label single arm post-market study where the purpose is to evaluate the effectiveness and safety of the market approved Spinal Simplicity Minuteman G5 MIS Fusion Plate and bone graft material in patients with degenerative conditions of the lumbar spine resulting in chronic low back pain with lower extremity symptoms and concurrent neurogenic claudication. The indication for the device under study is degenerative conditions of the lumbar spine resulting in back pain with lower extremity symptoms and neurogenic claudication.

DETAILED DESCRIPTION:
Up to 150 subjects will be enrolled and treated at up to 20 study sites. Qualified subjects will be enrolled and treated with the Minuteman G5 Device. Subjects will be seen at 1-, 3-, 6- and 12-months following study treatment.

Key outcome assessments will include gait and balance testing performed using BioMech Lab sensor technology to capture and deliver three-dimensional patient motion data to a mobile device that instantly analyzes, distills, and quantifies the information. Patient reported outcome measures will also be collected to evaluate pain, quality of life and satisfaction. During the primary assessment at 12-months post-treatment subject will be offered a computerized topography (CT) scan to evaluate spinal fusion.

After completion of the Month 12 visit all subjects will be asked to complete annual visits through 5 years, which include collection of PROMs, safety review, and can be completed in person or remote.

ELIGIBILITY:
Inclusion Criteria

A subject must MEET ALL of the following inclusion criteria:

1. Be a candidate for Spinal Simplicity Minuteman G5 Fusion Plate device per labeled indication
2. Be willing and capable of giving written consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the subject's participation has been provided
3. Be willing and capable of subjective evaluation, read and understand written questionnaires, and read, understand the written informed consent
4. Be 18 years of age or older at the time of enrollment
5. Have been diagnosed with degenerative conditions of the lumbar spine resulting in chronic low back pain with lower extremity symptoms and concurrent neurogenic claudication
6. Received at least 3 months of non-operative or conservative treatment without significant benefit in the opinion of the Investigator
7. Be willing and able to comply with study-related requirements, procedures and visits
8. Be on a stable pain medication regimen, as determined by the Investigator, for at least 30 days prior to enrolling in this study.
9. Must disclose any unresolved major issues of secondary gain (e.g., social, financial, legal), as determined by the Investigator. Including being involved in an injury claim under current litigation or has a pending or approved worker's compensation claim. Subjects will not be excluded due to secondary gain, but it should be disclosed at Enrollment.

Exclusion Criteria

A subject must NOT MEET ANY of the following exclusion criteria:

1. Had previous spinal surgery at the level of intervention (e.g. lumbar fusion, discectomy, Laminectomy) MILD procedure is not considered an exclusion.
2. Patient physically unable to perform the Gait and/or Balance tests.
3. Current systemic infection or local infection increasing the risk of surgery
4. History of medications decreasing bone quality or soft tissue healing in the opinion of the Investigator
5. Grade II-V spondylolisthesis
6. Significant scoliosis with Cobb angle >10 degrees
7. Unremitting back pain in a spinal flexion position
8. Active systemic disease that may affect the welfare of the subject in the opinion of the Investigator
9. Be concurrently participating in another clinical drug and/or device study that may alter or confound the results of the assessment (investigational device, investigational drug, new indication for a device or drug, or additional testing beyond standard of care procedures) as determined by the investigator.
10. Vertebral osteoporosis or history of vertebral fracture
11. Be pregnant/ lactating or plan to become pregnant from study enrollment through 3 months post-operatively. (determined by urine testing unless female subject is surgical sterile or post-menopausal). If female, sexually active and childbearing age, subject must be willing to use a reliable form of birth control through the 3-month visit.
12. Malformation or dysplasia of spinous process
13. Severe osteoporosis with T score <-2.5 SD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Pain (Overall, Back and Leg) using NRS/numeric rating scale | Baseline and 1-, 3-, 6- and 12-months post implantation; annually out to five years.
  Overall pain, as well as back pain when standing/walking and leg pain when standing will be assessed using a numeric rating scale (NRS). The NRS is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Oswestry Disability Index (ODI) | Baseline and 1-, 3-, 6- and 12-months post implantation; annually out to five years.
  ODI is a self-reported questionnaire widely used to track changes in a patient's condition over time and evaluate the effectiveness of treatments for low back pain. The ODI consists of 10 sections, each addressing a specific aspect of daily functioning. A higher score indicates greater disability. The final score/index ranges from 0-100 scale. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
PROMIS 29 2.0 | Baseline and 1-, 3-, 6- and 12-months post implantation; annually out to five years.
  PROMIS-29 c2.0 is a set of standardized questions that measures 29 items across 7 domains of physical and mental health. PROMIS-29 profile assesses pain intensity using a single 0-10 numeric rating scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable. And seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. Each domain is scored on T-Score Scale ranging between 22.9- 81.6 with a mean of 50 and a standard deviation of 10.
Assessment of Motion using BioMech Lab testing equipment | Baseline and 1-, 3- and 12-months post implantation.
  A Primary Objective of this study is to collect real-world functional outcomes assessment of motion following treatment with the market-released Spinal Simplicity Minuteman G5 Device using BioMech Lab equipment to record gait and balance. The BioMech Lab motion analytics system will assess gait and balance via sensors placed before physical testing.
Zurich Classification Questionnaire (ZCQ) | Baseline and 1-, 3- 6- and 12-months post implantation; annually out to five years.
  The ZCQ Symptom Severity, Physical Function and Subject Satisfaction allows subjects to rate their symptoms, function or satisfaction on a scale based on their experience over the past week.
  Symptom Severity domain evaluates the intensity of symptoms such as pain and numbness. It comprises seven items, each rated on a scale from 1 to 5. Overall symptom score ranges from 7-49; with higher scores indicating more severe symptoms.
  Physical Function domain assesses the impact of symptoms on daily activities. It includes five items, scored on a 1 to 4 scale. Overall symptom score ranges from 5-20; where higher scores denote greater functional impairment.
  Subject Satisfaction domain measures patient satisfaction with treatment outcomes. It consists of six items, each rated from 1 to 4, with higher scores reflecting greater dissatisfaction. Overall Satisfaction ranges from 6-24: where higher scores denote greater dissatisfaction.

SECONDARY OUTCOMES:
Spinal Fusion Assessment based on review of Lumbar Computerized Tomography (CT) Scan | Collected at 12 months post implantation.
  The secondary objective is to assess spinal fusion at 12 months post-operative using a Fusion Assessment Scale provided by Spinal Simplicity based on review of Lumbar CT Scan.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hedman, PhD, Study Chair — Spinal Simplicity
Locations (6):
- United States (6):
  - Vista Clinical Research, Newnan, Georgia
  - Comprehensive Pain & Spine Specialists, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Nura Precision Pain Management, Edina, Minnesota
  - Pacific Sports & Spine, Eugene, Oregon
  - Spine & Nerve Center of the Virginias, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No
Patients will be deidentified with unique study ID. Any study will be anonymized.